CLINICAL TRIAL: NCT03339557
Title: Functional Outcome of Total Knee Replacement. Randomized Clinical Controlled Trial of Novel and Conventional Implants
Brief Title: Comparison of Three Knee Replacements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Coxa, Hospital for Joint Replacement (Other)
Responsible Party: Principal Investigator, Tero Irmola, orthopaedic surgeon, Coxa, Hospital for Joint Replacement
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R15053
Record Dates: First submitted 2017-11-07; First posted 2017-11-13 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Osteoarthritis, Knee; Arthroplasty; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients will be recruited from Coxa outpatient clinic according to inclusion and exclusion criteria. The participating orthopedic surgeons will recruit patients along their out-patient work. The indications for the surgical treatment in the study will follow the routine clinical guidelines of the hospital. When TKR surgery is decided, the eligible patients will be informed and those willing to participate will be randomized into one of the three implant groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will be operated upon using the implant allocated in randomization. Participants are blinded to the implant design used for their operation. Staff at the ward is also blinded. And the physiotherapists conducting the follow-up visits (at 2-3 months, 1 year and 2 years, i.e. the outcome assessors) are also blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- PFC Total Knee Replacement (Active Comparator): PFC, Conventional design Perioperative treatment will be carried out according to routine protocol of the hospital.
  Interventions: Device: NexGen; Device: Persona
- NexGen Total Knee Replacement (Active Comparator): NexGen, Conventional design Perioperative treatment will be carried out according to routine protocol of the hospital.
  Interventions: Device: Persona; Device: PFC
- Persona Total Knee Replacement (Active Comparator): Persona, Novel design Perioperative treatment will be carried out according to routine protocol of the hospital.
  Interventions: Device: NexGen; Device: PFC

INTERVENTIONS:
Device: NexGen — Comparing two conventional designs and one novel design
  Arms: PFC Total Knee Replacement; Persona Total Knee Replacement
Device: Persona — Comparing two conventional designs and one novel design
  Arms: NexGen Total Knee Replacement; PFC Total Knee Replacement
Device: PFC — Comparing two conventional designs and one novel design
  Arms: NexGen Total Knee Replacement; Persona Total Knee Replacement

SUMMARY:
The present randomized controlled trial is designed to compare one novel total knee replacement (TKR) design and two conventional TKR designs in terms of functional outcome. 80 patients will be randomized in each of the three arms (240 altogether).

DETAILED DESCRIPTION:
The study will compare the short-term functional outcome (at 2 years) of TKR performed with a novel TKR design (Persona , Zimmer, Warsaw, IN, USA) against TKRs performed with two conventional designs (PFC, DePuy, Warsaw, IN, USA and Nexgen, Zimmer, Warsaw, IN, USA).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total knee replacement surgery for primary osteoarthritis
* no previous open major surgery in the joint ( e.g. osteotomy)
* unilateral operative treatment, with no plans for surgical treatment of the contralateral knee in the near future
* patients living in the local hospital district (Pirkanmaa Hospital District)
* Kellgren-Lawrence grade 3-4 knee osteoarthritis in plain radiographs

Exclusion Criteria:

* Unwilling to provide informed consent
* > 15 degrees varus or valgus, or >15 degree fixed flexion deformity
* predominantly patellofemoral osteoarthritis
* Physical, emotional or neurological conditions that would compromise the patient´s compliance with postoperative rehabilitation and follow-up (e.g. drug or alcohol abuse, serious mental illness, general neurological conditions such as Parkinson, MS, etc.)

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in patient reported outcome measures scores (PROMs), Functional improvement | preoperative, postoperative at 2-3 months, at 1 year and at 2 years
  Oxford Knee Score (OKS)

SECONDARY OUTCOMES:
Changes in PROMs, Functional improvement | preoperative, postoperative at 2-3 months, at 1 year and at 2 years
  Forgotten Joint Score (FJS)
Changes in health-related quality of life (HRQoL) | preoperative, postoperative at 2-3 months, at 1 year and at 2 years
  15D
Changes in activity rating scale | preoperative, postoperative at 2-3 months, at 1 year and at 2 years
  UCLA activity score
Changes in pain scale measurement | preoperative, postoperative at 2-3 months, at 1 year and at 2 years
  VAS pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Tero Irmola, MD, Principal Investigator — Coxa, Hospital for Joint Replacement
Locations (1):
- Coxa, Hospital for Joint Replacement, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ethgen O, Bruyere O, Richy F, Dardennes C, Reginster JY. Health-related quality of life in total hip and total knee arthroplasty. A qualitative and systematic review of the literature. J Bone Joint Surg Am. 2004 May;86(5):963-74. doi: 10.2106/00004623-200405000-00012. PMID 15118039
- [Background] Rasanen P, Paavolainen P, Sintonen H, Koivisto AM, Blom M, Ryynanen OP, Roine RP. Effectiveness of hip or knee replacement surgery in terms of quality-adjusted life years and costs. Acta Orthop. 2007 Feb;78(1):108-15. doi: 10.1080/17453670610013501. PMID 17453401
- [Background] Jenkins PJ, Clement ND, Hamilton DF, Gaston P, Patton JT, Howie CR. Predicting the cost-effectiveness of total hip and knee replacement: a health economic analysis. Bone Joint J. 2013 Jan;95-B(1):115-21. doi: 10.1302/0301-620X.95B1.29835. PMID 23307684
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Scott CE, Howie CR, MacDonald D, Biant LC. Predicting dissatisfaction following total knee replacement: a prospective study of 1217 patients. J Bone Joint Surg Br. 2010 Sep;92(9):1253-8. doi: 10.1302/0301-620X.92B9.24394. PMID 20798443
- [Background] Beswick AD, Wylde V, Gooberman-Hill R, Blom A, Dieppe P. What proportion of patients report long-term pain after total hip or knee replacement for osteoarthritis? A systematic review of prospective studies in unselected patients. BMJ Open. 2012 Feb 22;2(1):e000435. doi: 10.1136/bmjopen-2011-000435. Print 2012. PMID 22357571
- [Background] Giesinger K, Hamilton DF, Jost B, Holzner B, Giesinger JM. Comparative responsiveness of outcome measures for total knee arthroplasty. Osteoarthritis Cartilage. 2014 Feb;22(2):184-9. doi: 10.1016/j.joca.2013.11.001. Epub 2013 Nov 18. PMID 24262431
- [Background] Hamilton DF, Gaston P, Simpson AH. Is patient reporting of physical function accurate following total knee replacement? J Bone Joint Surg Br. 2012 Nov;94(11):1506-10. doi: 10.1302/0301-620X.94B11.30081. PMID 23109630
- [Background] Behrend H, Giesinger K, Giesinger JM, Kuster MS. The "forgotten joint" as the ultimate goal in joint arthroplasty: validation of a new patient-reported outcome measure. J Arthroplasty. 2012 Mar;27(3):430-436.e1. doi: 10.1016/j.arth.2011.06.035. Epub 2011 Oct 13. PMID 22000572
- [Background] Thienpont E, Opsomer G, Koninckx A, Houssiau F. Joint awareness in different types of knee arthroplasty evaluated with the Forgotten Joint score. J Arthroplasty. 2014 Jan;29(1):48-51. doi: 10.1016/j.arth.2013.04.024. Epub 2013 May 18. PMID 23688851
- [Background] Klit J, Jacobsen S, Rosenlund S, Sonne-Holm S, Troelsen A. Total knee arthroplasty in younger patients evaluated by alternative outcome measures. J Arthroplasty. 2014 May;29(5):912-7. doi: 10.1016/j.arth.2013.09.035. Epub 2013 Oct 1. PMID 24269097
- [Background] Grosu I, Lavand'homme P, Thienpont E. Pain after knee arthroplasty: an unresolved issue. Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1744-58. doi: 10.1007/s00167-013-2750-2. Epub 2013 Nov 8. PMID 24201900
- [Background] Singh JA, Gabriel S, Lewallen D. The impact of gender, age, and preoperative pain severity on pain after TKA. Clin Orthop Relat Res. 2008 Nov;466(11):2717-23. doi: 10.1007/s11999-008-0399-9. Epub 2008 Aug 5. PMID 18679762
- [Background] Perez-Prieto D, Gil-Gonzalez S, Pelfort X, Leal-Blanquet J, Puig-Verdie L, Hinarejos P. Influence of depression on total knee arthroplasty outcomes. J Arthroplasty. 2014 Jan;29(1):44-7. doi: 10.1016/j.arth.2013.04.030. Epub 2013 May 20. PMID 23702267
- [Background] Hanusch BC, O'Connor DB, Ions P, Scott A, Gregg PJ. Effects of psychological distress and perceptions of illness on recovery from total knee replacement. Bone Joint J. 2014 Feb;96-B(2):210-6. doi: 10.1302/0301-620X.96B2.31136. PMID 24493186
- [Background] Dowsey MM, Nikpour M, Dieppe P, Choong PF. Associations between pre-operative radiographic osteoarthritis severity and pain and function after total hip replacement : Radiographic OA severity predicts function after THR. Clin Rheumatol. 2016 Jan;35(1):183-9. doi: 10.1007/s10067-014-2808-7. Epub 2014 Oct 24. PMID 25339125
- [Background] Keurentjes JC, Fiocco M, So-Osman C, Onstenk R, Koopman-Van Gemert AW, Poll RG, Kroon HM, Vliet Vlieland TP, Nelissen RG. Patients with severe radiographic osteoarthritis have a better prognosis in physical functioning after hip and knee replacement: a cohort-study. PLoS One. 2013;8(4):e59500. doi: 10.1371/journal.pone.0059500. Epub 2013 Apr 3. PMID 23573200
- [Background] Berend KR, Lombardi AV Jr, Adams JB. Which total knee replacement implant should I pick? Correcting the pathology: the role of knee bearing designs. Bone Joint J. 2013 Nov;95-B(11 Suppl A):129-32. doi: 10.1302/0301-620X.95B11.32835. PMID 24187370
- [Background] van der Voort P, Pijls BG, Nouta KA, Valstar ER, Jacobs WC, Nelissen RG. A systematic review and meta-regression of mobile-bearing versus fixed-bearing total knee replacement in 41 studies. Bone Joint J. 2013 Sep;95-B(9):1209-16. doi: 10.1302/0301-620X.95B9.30386. PMID 23997134
- [Background] Becker R, Hirschmann MT, Karlsson J. Does implant design and surgical technique improve the clinical outcome in total knee arthroplasty? Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1716-8. doi: 10.1007/s00167-014-3145-8. No abstract available. PMID 24981991
- [Background] Nunley RM, Nam D, Berend KR, Lombardi AV, Dennis DA, Della Valle CJ, Barrack RL. New total knee arthroplasty designs: do young patients notice? Clin Orthop Relat Res. 2015 Jan;473(1):101-8. doi: 10.1007/s11999-014-3713-8. PMID 24903823
- [Background] Baker PN, Deehan DJ, Lees D, Jameson S, Avery PJ, Gregg PJ, Reed MR. The effect of surgical factors on early patient-reported outcome measures (PROMS) following total knee replacement. J Bone Joint Surg Br. 2012 Aug;94(8):1058-66. doi: 10.1302/0301-620X.94B8.28786. PMID 22844046
- [Background] Piepers MJ, van Hove RP, van den Bekerom MP, Nolte PA. Do refinements to original designs improve outcome of total knee replacement? A retrospective cohort study. J Orthop Surg Res. 2014 Feb 6;9:7. doi: 10.1186/1749-799X-9-7. PMID 24502700
- [Background] Pritchett JW. Patients prefer a bicruciate-retaining or the medial pivot total knee prosthesis. J Arthroplasty. 2011 Feb;26(2):224-8. doi: 10.1016/j.arth.2010.02.012. Epub 2010 Oct 6. PMID 20932707
- [Derived] Irmola T, Kangas J, Eskelinen A, Niemelainen M, Huhtala H, Mattila VM, Moilanen T. Functional outcome of total knee replacement: a study protocol for a prospective, double-blinded, parallel-group randomized, clinical controlled trial of novel, personalized and conventional implants. BMC Musculoskelet Disord. 2019 Oct 12;20(1):443. doi: 10.1186/s12891-019-2830-7. PMID 31604440